CLINICAL TRIAL: NCT00816075
Title: The Efficacy of Distilled Water vs Mitomycin C as a Single Dose Immediate Instillation After Transurethral Resection of Intermediate Risk, Recurrent Superficial Bladder Cancer
Brief Title: Efficacy of Distilled Water Versus Mitomycin C on Preventing Recurrences of Bladder Cancer After Transurethral Resection
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Zafer Kozacioglu, Bozyaka Training and Research Hospital Urology Clinic
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: URO-DW-1971
Record Dates: First submitted 2008-12-30; First posted 2008-12-31 (Estimated); Last update posted 2009-02-17 (Estimated); Status verified 2009-02

CONDITIONS: Recurrent Superficial Bladder Cancer; Distilled Water
Keywords: distilled water; recurrent; bladder; mitomycin
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Recurrence

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1, Distilled water (Experimental): the group of patients with superficial bladder cancer in the intermediate risk group who had their first recurrence after 6 months from the initial TUR. We plan to administer 200 ml of distilled water as immediate instillation for 2 hours
  Interventions: Drug: distilled water

INTERVENTIONS:
Drug: distilled water — we plan to administer 200ml of distilled water after TUR of the tumor and block the catheter for 2 hours

SUMMARY:
The purpose of this study is to compare and evaluate the efficacy of distilled water vs Mitomycin C on preventing the recurrences of intermediate risk group recurrent superficial bladder cancer administered as a single dose immediate instillation after complete Transurethral Resection(TUR) of the tumor.

DETAILED DESCRIPTION:
We plan to administer 200ml of distilled water as a single peroperative instillation and block the catheter for 2 hours to our eligible recurrent superficial bladder cancer patients who were in our follow-up schedule since 2002.

We plan to look over the histories of the same patients in terms of the pathologies, recurrence patterns, the presence of peroperative intracavitary therapy after their previous TURs for recurrences.

So we shall compare the effectiveness of MMC and distilled water on reducing the recurrences over the same patient pool.

The patients will be scheduled for a follow-up program after TUR as;

* cystoscopy
* urine cytology
* bladder wash cytology for the probability of recurrence for 2 years to see if there is any difference in the recurrence patterns after instillation with distilled water vs MMC.

ELIGIBILITY:
Inclusion Criteria:

* pathologic finding of superficial bladder cancer within the intermediate risk group
* recurred after 6 months from the primary tumor
* those patients who were included in our follow-up program since 2002 and whose records could be obtained.

Exclusion Criteria:

* carcinoma in situ
* any form of intracavitary maintenance therapy
* any form of bladder cancer other than transitional cell type

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-01 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
tumor recurrence by cystoscopic examination, urine and bladder wash cytology | within two years after instillation

CONTACTS AND LOCATIONS:
Overall Officials: Zafer Kozacioglu, MD, Principal Investigator — Bozyaka Trainig and Research Hospital Urology Clinic; Murat Arslan, MD, Study Chair — Bozyaka Training and Research Hospital Urology Clinic; Tansu Degirmenci, MD, Study Chair — Bozyaka Training and Research Hospital Urology Clinic; Fatih Duz, MD, Study Chair — Bozyaka Training and Research Hospital Urology Clinic; Ali R Ayder, MD, Study Director — Bozyaka Training and Research Hospital Urology Clinic; Nukhet Eliyatkin, MD, Study Chair — Bozyaka Training and Research Hospital Pathology Clinic
Locations (1):
- Bozyaka Training and Research Hospital Urology Clinic, Izmir, Turkey (Türkiye)